CLINICAL TRIAL: NCT03293108
Title: A Phase III, Randomized, Two-armed, Parallel, Double-blind, Active-controlled, Non-inferiority Clinical Trial to Determine the Non-inferior Therapeutic Efficacy and Safety Between Arylia (60 mg, Denosumab, Produced by AryoGen Pharmed) Compared With Prolia® (60 mg, Denosumab, the Reference Drug, Produced by Amgen Company) in the Improvement of Bone Mineral Densitometry (BMD) Among Osteoporotic Postmenopausal Women
Brief Title: Comparing Efficacy and Safety of AryoGen Pharmed Biosimilar Denosumab 60 mg (Arylia) Versus Prolia® in Improvement of Bone Mineral Densitometry (BMD) Among Osteoporotic Postmenopausal Women
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: AryoGen Pharmed Co. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DEN.ARY.AJ.95 (III)
Record Dates: First submitted 2017-09-19; First posted 2017-09-26 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Osteoporosis
Keywords: Osteoporosis; Denosumab
MeSH Terms: conditions — Osteoporosis | interventions — Denosumab; Calcium; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AryoGen Pharmed Denosumab (Experimental): Arylia (Denosumab Prefilled Syringe produced by AryoGen Pharmed) 60 mg/1 ml in a prefilled syringe.
  Denosumab 60 mg is subcutaneously administered to osteoporotic patients at baseline, month 6 and month 12. Along with, all women will receive daily supplements containing at least 1000 mg of elemental calcium (divided into two doses) and at least 400 IU vitamin D daily during 18 months of the study.
  Interventions: Drug: Denosumab; Dietary Supplement: calcium; Dietary Supplement: vitamin D
- Amgen Denosumab (Active Comparator): Prolia® (Denosumab Prefilled Syringe produced by Amgen) 60 mg/1 ml in a prefilled syringe.
  Denosumab 60 mg is subcutaneously administered to osteoporotic patients at baseline, month 6 and month 12. Along with, all women will receive daily supplements containing at least 1000 mg of elemental calcium (divided into two doses) and at least 400 IU vitamin D daily during 18 months of the study.
  Interventions: Drug: Denosumab; Dietary Supplement: calcium; Dietary Supplement: vitamin D

INTERVENTIONS:
Drug: Denosumab — Denosumab 60 mg is subcutaneously administered to osteoporotic patients at baseline, month 6 and month 12.
Dietary Supplement: calcium — All women will receive daily supplements containing at least 1000 mg of elemental calcium (divided in two doses), during 18 month of the study.
Dietary Supplement: vitamin D — All women will receive daily supplements containing at least 400 IU vitamin D daily during 18 month of the study.

SUMMARY:
The purpose of this study is to compare the efficacy and safety of Denosumab 60 mg produced by AryoGen Pharmed and Amgen Denosumab 60 mg among osteoporotic postmenopausal women. Postmenopausal women diagnosed with osteoporosis according to their Bone mineral density result (BMD), aged between 45 to 75 are included in this trial. This is a Phase III, randomized, two armed, double-blind, parallel, active-controlled,non-inferiority clinical trial. The eligible patients are randomized in a 1:1 ratio to receive Arylia or Prolia® subcutaneous injections, at the beginning of the trial and every 6 months at month 6 and 12, in an 18-month study period. Along with, all women will receive daily supplements containing at least 1000 mg of elemental calcium (divided into two doses) and at least 400 IU vitamin D daily during 18 months of the study.

The primary objective of this study is to assess non-inferiority of test- Denosumab 60 mg (Arylia) to the reference Denosumab 60 mg (Prolia®) in terms of efficacy among osteoporotic postmenopausal women.

The secondary objectives of this study are:

To further compare efficacy of test- Denosumab 60 mg to reference Denosumab 60 mg; To assess the safety of test- Denosumab 60 mg compared to reference Denosumab 60 mg.

DETAILED DESCRIPTION:
The purpose of this study is to compare the efficacy and safety of Denosumab 60 mg produced by AryoGen Pharmed and Amgen Denosumab 60 mg among osteoporotic postmenopausal women. Postmenopausal women diagnosed with osteoporosis according to their Bone mineral density result (BMD) and aged between 45 to 75 are included in this trial. This is a Phase III, randomized, two armed, double-blind, parallel, active-controlled,non-inferiority clinical trial. Visits are going to be conducted at screening, 0, 1, 3, 6, 9, 12, 15 and 18 months.

After signing the written informed consent, patients are randomized in a 1:1 ratio to receive Arylia or Prolia® subcutaneous injections, at the beginning of the trial and every 6 months at month 6 and 12, in an 18-month study period. Along with, all women will receive daily supplements containing at least 1000 mg of elemental calcium (divided into two doses) and at least 400 IU vitamin D daily during 18 months of the study.

The primary objective of this study is to assess percentage change from baseline in BMD at the lumbar spine (L1-L4), femoral neck and total hip by dual-energy x-ray absorptiometry to 18 months of the study, and compare it between two treatment groups.

The second objectives of this study are to assess the followings between treatment groups:

* The incidence of new vertebral fracture;
* Evolution of biochemical markers of bone metabolism at baseline, first month and afterward every 3 months from baseline.
* Comparing adverse events;
* Comparing immunogenicity of two products.

Before initiation, the trial is reviewed by food and drug administration of Iran. The protocol, electronic case report form (eCRF), information for patients and informed consent forms are submitted to the ethics committees responsible for review and approval purposes, according to national regulatory guidelines.

Sample size:

172 patients will be equally (1:1) divided into intervention arms for achieving 80% power in order to determine non-inferiority using a one-sided, independent sample t-test. Efficacy of Prolia® in comparison with placebo for lumbar spine BMD improvement in previous studies is reported 7.1%. The margin of non-inferiority is 1.78. The true difference between the means is assumed to be 0.000. The significance level (alpha) of the test is 0.025. The data are drawn from populations with standard deviations of 4.116 and 4.116. However, we have calculated that 190 patients should enter the study, by considering that there might be 10% drop-outs of participants during the trial.

Blinding:

To prevent the influence of knowing intervention group on study conclusion, the subjects and those who assess the study outcomes will be unaware of the state of the patient with regard to receiving the test drug or reference drug.

For this purpose, subjects and administrator of the drug will be blinded by using a similar masked prefilled syringes. All drugs packages will be identified by unique numbers.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women aged between 45 up to 75;
* Bone mineral density T score at the lumbar spine (L1-L4), femoral neck or total hip should be equal or less than -2.5 and equal or more than -4. (-4 ≤ T score ≤-2.5); or patients with high risk of fracture on the basis of FRAX criteria which according to osteoporosis treatment guidelines, need medicinal treatment.
* Ability to comprehend and willingness to sign the Informed Consent Form for this study;
* Signed informed consent with full knowledge and mental health.

Exclusion Criteria:

* Lack of consent for being in the trial and not complying with an 18-months follow-up;
* Having hypersensitivity to denosumab or any component in the formulation (excipients include acetic acid, sorbitol, polysorbate 20, sodium hydroxide, water for injections);
* Malabsorption syndrome;
* History of thyroid surgery, parathyroid surgery or intestinal resection which has been caused malabsorption.
* Patient with CKD stage 4 and 5 should be exclude (GFR <30cc/min)
* Level of serum 25-(OH) vitamin D less than 20 ng/ml; (If vitamin deficiency has been corrected, and two tests show the level above 20 ng/ml within a month, the patient can be enrolled.)
* Pre-existing hypocalcemia (Albumin-adjusted serum calcium level less than 8 mg/dl in fasting specimens) which is uncorrectable;
* Untreated hypercalciuria (>250 mg/24h) and hypocalciuria (<100 mg/24h). If urine calcium level of patient is less than 100 mg per 24 hours and by vitamin D treatment the problem has been solved or if urine calcium level of patient is greater than 250 mg per 24 hours, but PTH is normal, the patient can be enrolled.
* Presence of osteonecrosis of jaw (ONJ) risk factors including a diagnosis of cancer, poor oral hygiene, periodontal and/or dental diseases, having dentures; and comorbid disorders (anemia (hemoglobin level less than 11 g/dl, if it is corrected, patient can enter the study), history of diseases with coagulopathy, oral and dental infection);
* Malignancy;
* Having severe and active infections; (Severe infection is a difficult treated infection, like diabetic foot infection, but if the infection is treatable, after treatment, the patient can be enrolled.)
* Being bed rest (for 2 weeks during the past 3 months)
* A case in which the patient cannot take 1000 mg oral elemental calcium per day; (as supplement)
* A case in which bone mineral density could not be accurately measured;
* Conditions that influence bone metabolism, including hyperparathyroidism or hypoparathyroidism, hyperthyroidism or hypothyroidism, hypocalcemia, inflammatory rheumatologic diseases such as rheumatoid arthritis, Paget's disease of bone, osteomalacia that is resistant to therapy (definition of resistant to therapy: not being responder to 1-month administration of vitamin D).
* Patients will be excluded if they have one severe or more than 2 moderate vertebral fractures. (Severe fracture is defined as more than 50 percent vertebral height loss and moderate fracture is defined as 25-50 percent vertebral height loss).
* Use of injectable bisphosphonates within the previous 12 months;
* Use of oral bisphosphonates within the previous 3 months;
* History of severe skeletal pain with bisphosphonates;
* Use of parathyroid hormone or its derivatives, systemic hormone-replacement therapy, selective estrogen-receptor modulator, calcitonin, or calcitriol within 6 weeks before study enrollment.
* Use of corticosteroids (>5 mg/prednisone daily or equivalent for ≥ 3months), in the past 3 months and more.
* Use of heparin (more than 20,000 international units/day for 6 months and longer), in the past 6 months and more.
* Patient that is possible to be administrated corticosteroids (>5 mg/prednisone daily or equivalent for ≥ 3months) or heparin (more than 20,000 international units/day for 6 months and longer) in the 18 month of the study, because of her chronic disease(s) such as allergy, asthma, coagulation disorders, should be excluded.

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2017-04-29 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
BMD percentage change from baseline at lumbar spine (L1-L4), femoral neck and total hip. | Baseline and at 18 months.
  Percentage change from baseline in BMD at lumbar spine (L1-L4), femoral neck and total hip by dual-energy x-ray absorptiometry to 18 months of the study, and compare between two groups.

SECONDARY OUTCOMES:
The incidence of new vertebral fracture. | Baseline and at 18 months
  The incidence of new vertebral fracture assessed by Lateral spine X-ray radiography (T4-L4) at baseline then at 18 months, and compare between two groups.
Evolution of biochemical markers of bone metabolism. | Baseline,at month 1,at month 3,at month 6,at month 9, at month 12, at month 15 and at month 18.
  Evolution of biochemical markers of bone metabolism at baseline, first month and afterwards every 3 months from baseline, and compare between two groups.
Comparing adverse events between two products. | baseline,at month 1,at month 3,at month 6,at month 9,at month 12, at month 15 and at month 18.
  Evaluation of the following parameters at each visit including 0, 1, 3, 6, 9, 12, 15 and 18 months, and compare between two groups.
  * Adverse events (AEs), Adverse drug reactions (ADR)
  * Changes in physical examination findings
  * Changes in vital signs
  * Clinical laboratory testing for systemic safety, including liver function, renal function, complete blood count, and clinical chemistries.
Comparing immunogenicity between two products. | Baseline,at month 6,at month 12 and at month 18.
  Evaluation of immunogenicity at visit 0, 6, 12 and 18 months for both arms, and compare between two groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Rheumatology Center of Iran, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lim SY, Bolster MB. Current approaches to osteoporosis treatment. Curr Opin Rheumatol. 2015 May;27(3):216-24. doi: 10.1097/BOR.0000000000000169. PMID 25760281
- [Background] Drake MT, Clarke BL, Lewiecki EM. The Pathophysiology and Treatment of Osteoporosis. Clin Ther. 2015 Aug;37(8):1837-50. doi: 10.1016/j.clinthera.2015.06.006. Epub 2015 Jul 7. PMID 26163201
- [Background] Cosman F, de Beur SJ, LeBoff MS, Lewiecki EM, Tanner B, Randall S, Lindsay R; National Osteoporosis Foundation. Clinician's Guide to Prevention and Treatment of Osteoporosis. Osteoporos Int. 2014 Oct;25(10):2359-81. doi: 10.1007/s00198-014-2794-2. Epub 2014 Aug 15. PMID 25182228
- [Background] Cairoli E, Eller-Vainicher C, Chiodini I. Update on denosumab in the management of postmenopausal osteoporosis: patient preference and adherence. Int J Womens Health. 2015 Oct 13;7:833-9. doi: 10.2147/IJWH.S75681. eCollection 2015. PMID 26508890
- [Background] Diedhiou D, Cuny T, Sarr A, Norou Diop S, Klein M, Weryha G. Efficacy and safety of denosumab for the treatment of osteoporosis: A systematic review. Ann Endocrinol (Paris). 2015 Dec;76(6):650-7. doi: 10.1016/j.ando.2015.10.009. Epub 2015 Nov 27. PMID 26639186
- [Background] Herrero S, Pico Y. Treatments for post-menopausal osteoporotic women, what's new? How can we manage long-term treatment? Eur J Pharmacol. 2016 May 15;779:8-21. doi: 10.1016/j.ejphar.2016.02.053. Epub 2016 Feb 26. PMID 26923729
- [Background] Black DM, Rosen CJ. Clinical Practice. Postmenopausal Osteoporosis. N Engl J Med. 2016 Jan 21;374(3):254-62. doi: 10.1056/NEJMcp1513724. PMID 26789873
- [Background] Cummings SR, San Martin J, McClung MR, Siris ES, Eastell R, Reid IR, Delmas P, Zoog HB, Austin M, Wang A, Kutilek S, Adami S, Zanchetta J, Libanati C, Siddhanti S, Christiansen C; FREEDOM Trial. Denosumab for prevention of fractures in postmenopausal women with osteoporosis. N Engl J Med. 2009 Aug 20;361(8):756-65. doi: 10.1056/NEJMoa0809493. Epub 2009 Aug 11. PMID 19671655
- [Background] McClung MR, Lewiecki EM, Cohen SB, Bolognese MA, Woodson GC, Moffett AH, Peacock M, Miller PD, Lederman SN, Chesnut CH, Lain D, Kivitz AJ, Holloway DL, Zhang C, Peterson MC, Bekker PJ; AMG 162 Bone Loss Study Group. Denosumab in postmenopausal women with low bone mineral density. N Engl J Med. 2006 Feb 23;354(8):821-31. doi: 10.1056/NEJMoa044459. PMID 16495394
- [Background] Brown JP, Prince RL, Deal C, Recker RR, Kiel DP, de Gregorio LH, Hadji P, Hofbauer LC, Alvaro-Gracia JM, Wang H, Austin M, Wagman RB, Newmark R, Libanati C, San Martin J, Bone HG. Comparison of the effect of denosumab and alendronate on BMD and biochemical markers of bone turnover in postmenopausal women with low bone mass: a randomized, blinded, phase 3 trial. J Bone Miner Res. 2009 Jan;24(1):153-61. doi: 10.1359/jbmr.0809010. PMID 18767928
- [Background] Gu HF, Gu LJ, Wu Y, Zhao XH, Zhang Q, Xu ZR, Yang YM. Efficacy and Safety of Denosumab in Postmenopausal Women With Osteoporosis: A Meta-Analysis. Medicine (Baltimore). 2015 Nov;94(44):e1674. doi: 10.1097/MD.0000000000001674. PMID 26554766
- [Background] Bone HG, Bolognese MA, Yuen CK, Kendler DL, Wang H, Liu Y, San Martin J. Effects of denosumab on bone mineral density and bone turnover in postmenopausal women. J Clin Endocrinol Metab. 2008 Jun;93(6):2149-57. doi: 10.1210/jc.2007-2814. Epub 2008 Apr 1. PMID 18381571
- [Derived] Jamshidi A, Vojdanian M, Soroush M, Akbarian M, Aghaei M, Hajiabbasi A, Mirfeizi Z, Khabbazi A, Alishiri G, Haghighi A, Salimzadeh A, Karimzadeh H, Shirani F, Fard MRH, Nazarinia M, Soroosh S, Anjidani N, Gharibdoost F. Efficacy and safety of the biosimilar denosumab candidate (Arylia) compared to the reference product (Prolia(R)) in postmenopausal osteoporosis: a phase III, randomized, two-armed, double-blind, parallel, active-controlled, and noninferiority clinical trial. Arthritis Res Ther. 2022 Jun 30;24(1):161. doi: 10.1186/s13075-022-02840-8. PMID 35773713